CLINICAL TRIAL: NCT05585034
Title: A Phase 1, First-in-Human, Dose-Finding and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Activity of XmAb®808 in Combination With Pembrolizumab in Selected Advanced Solid Tumors
Brief Title: Phase 1, First-in-human, Dose-finding and Expansion Study to Evaluate XmAb®808 in Combination With Pembrolizumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb808-01
Record Dates: First submitted 2022-10-11; First posted 2022-10-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Melanoma Excluding Uveal Melanoma; Non-small Cell Lung Cancer, Squamous or Non-squamous; Urothelial Carcinoma; Renal Cell Carcinoma, Clear Cell; Castration-resistant Prostate Cancer; Ovarian Cancer, Epithelial; TNBC - Triple-Negative Breast Cancer; Colorectal Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Triple Negative Breast Neoplasms; Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation and Expansion XmAb®808 administered in combination with pembrolizumab (Experimental): XmAb®808 in combination with pembrolizumab
  Interventions: Biological: XmAb®808; Biological: Keytruda® (pembrolizumab)

INTERVENTIONS:
Biological: XmAb®808 — Monoclonal bispecific antibody
Biological: Keytruda® (pembrolizumab) — Monoclonal antibody

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of intravenous (IV) administration of XmAb808 in combination with pembrolizumab in subjects with selected advanced solid tumors and to identify the minimum safe and biologically effective/recommended dose (RD) and schedule for XmAb808.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, first-in-human (FIH), multiple-dose, dose escalation study with cohort expansion at the RD, designed to evaluate the safety and tolerability of XmAb808 in combination with pembrolizumab. This study will be conducted in 2 parts: Part A (dose escalation) and Part B (cohort expansion).

ELIGIBILITY:
Key Inclusion Criteria:

* Part A: Histologically confirmed advanced/metastatic castration-resistant prostate adenocarcinoma, epithelial ovarian cancer, head and neck squamous cell carcinoma, non-small cell lung cancer, urothelial carcinoma, melanoma, renal cell carcinoma, triple-negative breast cancer, or colorectal cancer that has progressed on standard therapies
* Part B: Histologically confirmed advanced/metastatic castration-resistant prostate cancer that is PD1-naïve; head and neck squamous cell carcinoma that is PD1-naïve or has progressed on prior PD1 therapy; or melanoma that is PD1-naïve or has progressed on prior PD1 therapy
* Measurable disease by RECIST 1.1; subjects with prostate cancer who have evaluable disease according to PCWG3 criteria may enroll
* Life expectancy > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Key Exclusion Criteria:

* Subjects currently receiving other anticancer therapies
* Any prior treatment with an investigational agent targeting CD28
* History of a life-threatening adverse event related to prior immunotherapy
* Known active central nervous system involvement by malignant disease. Subjects with previously treated brain metastases may participate provided they are radiologically and clinically stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 5 years
  Safety and tolerability as assessed by incidence of TEAEs, including clinically significant changes in safety laboratory tests and clinical findings
Incidence of dose-limiting toxicities (DLTs) | 49 days
  Safety and tolerability as assessed by incidence of DLTs and all available data which will be used to determine the optimal dose regimen

SECONDARY OUTCOMES:
Measurement of Cmax | Through study completion, Up to 5 years
  Peak plasma concentration (Cmax)
Measurement of AUCtau | Through study completion, Up to 5 years
  Area under the plasma concentration versus time curve (AUCtau)
Objective Response Rate | Through study completion, Up to 5 years
  Objective response rate by RECIST 1.1 assessment of CT/MRI imaging, as modified by PCWG3 for participants with prostate cancer
Progression-free Survival | Through study completion, Up to 5 years
  Progression-free survival by RECIST 1.1 assessment of CT/MRI imaging, as modified by PCWG3 for participants with prostate cancer
Duration of Response | Through study completion, Up to 5 years
  Duration of Response by RECIST 1.1 assessment of CT/MRI imaging, as modified by PCWG3 for participants with prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mira Kistler, MD, Study Director — Xencor, Inc.
Locations (12):
- United States (12):
  - UCLA Hematology/Oncology, Los Angeles, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Columbia University Irvine Medical Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Froedtert Hospital & The Medical College of Wisconsin, Milwaukee, Wisconsin